CLINICAL TRIAL: NCT01893385
Title: Impact of Vitamin D Supplementation on Immune Functions: Study in Subjects Aged Over 65 Years Vaccinated Against Influenza
Brief Title: Vitamin D Supplementation and the Immune Response
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0160; 2012-005658-52
Record Dates: First submitted 2013-06-25; First posted 2013-07-09 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: D Vitamin Deficiency Patients
Keywords: vitamin D; supplementation; immunocompetente cells, immune system; influenza vaccine; elderly
MeSH Terms: conditions — Influenza, Human | interventions — Vitamin D; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- vitamin D (Experimental): The entire project will collect new information on the merits of the use of vitamin D in aging. A better knowledge of mechanisms involved and the impact of aging on them is a necessary prerequisite the definition of a new strategy using this drug in the elderly particularly fragile in order to improve its autonomy. This definition seems a sociological interest obvious economic knowing the current aging population and its impact future of our health system
  Interventions: Drug: Vitamin D (drug)
- INTANZA 15 (Other): The entire project will collect new information on the merits of the use of vitamin D in aging. A better knowledge of mechanisms involved and the impact of aging on them is a necessary prerequisite the definition of a new strategy using this drug in the elderly particularly fragile in order to improve its autonomy. This definition seems a sociological interest obvious economic knowing the current aging population and its impact future of our health system
  Interventions: Drug: Vitamin D (drug)

INTERVENTIONS:
Drug: Vitamin D (drug)

SUMMARY:
The main objective is to assess the variation in plasma levels of cathelicidin before and after influenza vaccination.

All bibliographic data suggests that supplementation vitamin D in the elderly often deficient in this vitamin may have a double interest:

* By induction of cathelicidin, assist in anti-infective response in particular to the influenza virus
* The normalization of vitamin D status, promote the return to an appropriate immune response limiting excess inflammation and improving capacity to respond.

The entire project will collect new information on the merits of the use of vitamin D in aging. A better knowledge of mechanisms involved and the impact of aging on them is a necessary prerequisite the definition of a new strategy using this drug in the elderly particularly fragile in order to improve its autonomy. This definition seems a sociological interest obvious economic knowing the current aging population and its impact future of our health system.

DETAILED DESCRIPTION:
CONDUCT OF THE STUDY:

Visit 1: selection of subjects (CPC / CIC-Inserm CIC501)

* Medical Examination, clinical examination, explanation of the protocol and collection of written consent,
* Collection of anthropometric data measured size and not declarative weight form examination, measurement of current weight, BMI, waist circumference measurement.
* Food Survey.
* Fasting blood sampling: for dosing of vitamin D, cathelicidin, exploration of immunocompetent cells, calcium, phosphorus, urea and creatinine.

Visit 2: randomization (CPC / CIC-Inserm CIC501)

* Fasting blood sampling: for dosing of vitamin D, cathelicidin, and the serum calcium, phosphorus, urea and creatinine.
* Exploration of immune cells in patients deficient in vitamin D (molecular and cellular analyzes).

Start of vitamin D supplementation or placebo

* Subjects with vitamin D levels <30ng/mL will be randomized into two groups:

  * Arm receiving vitamin D (BS).
  * Arm receiving placebo (BC).
* It will be given to the patient 4 bulbs product (vitamin D or placebo) for supplementation for 2 months (1 / 15 days).

Call subjects at 4 weeks of vitamin supplementation / placebo to assess the clinical safety of the product, as well as compliance with the instructions of supplementation.

Visit 3: After seven weeks of vitamin supplementation / placebo (CPC / CIC-Inserm CIC501)

* Fasting blood assay for vitamin D and calcium collection.
* urinary dosage calcium. Visit 4: Month 2 (CPC / CIC-Inserm CIC501)
* Validation of laboratory measurements made by an independent medical M2 protocol.
* Delivery of products to test for the third month of vitamin supplementation / placebo.

For the placebo group given two bulbs for the third month placebo placebo supplementation.

For the VitD group: dose adjustment according to the following scheme:

* If [25(OH) D]> 75 ng / ml and / or calcium levels> 106 mg / ml and / or calcium excretion> 300 mg / l: presentation of two bulbs placebo.
* If [25(OH) D] <75 ng / ml and serum calcium <106 mg / ml and calcium excretion <300 mg / l: presentation of two ampoules of Vitamin D. Visit 5 - Month 3 vaccination INTANZA 15 ® (3 months after the start of supplementation)
* Recovery of boxes and empty ampoules of vitamin D.
* Evaluation of the clinical safety of vitamin D.
* Collection of anthropometric data: measurement of current weight and BMI,
* Fasting blood sampling: for dosing of vitamin D, cathelicidin, exploration of immunocompetent cells, calcium, phosphorus, urea and creatinine.
* Influenza serology, Visit 6 - Month 4: end of study
* Clinical examination with assessment of tolerability of vaccination and delivery of the form of reporting due to immunization and infectious complications side effects according to the criteria of toxicity CTCNCI Bethesda,
* Collection of anthropometric data: measurement of current weight, calculating the weight change,
* Fasting blood sampling: for dosing of vitamin D, cathelicidin, exploration of immunocompetent cells, calcium, phosphorus, urea and creatinine.
* Measurement of seroconversion, seroprotection, MGT antibodies following vaccination.

End of the study Removal of anonymity for physician investigators to propose a vitamin D the subjects who received placebo.

ELIGIBILITY:
Inclusion Criteria:

- Aged 65 or over subject,

* Subjects with a vitamin D levels below 30 ng / ml,
* Acceptance of vitamin D (100 000 IU of UVEDOSE ®)
* Acceptance of influenza vaccination with INTANZA15 ®
* Affiliation to a social security scheme
* The subject agrees not to change their eating habits

Exclusion Criteria:

* Liver disease: cirrhosis, chronic hepatitis.
* Renal impairment whatever degree
* Hypercalcemia (serum calcium> 2.6 mol / l)
* Hypo-or hyperparathyroidism history, history of renal colic.
* Disease / acute infection, moderate or severe (at the discretion of the investigator) on the day of vaccination or febrile illness (temperature ≥ 38 ° C). The subject should not be included in the study as his condition is not cured or her fever has not gone down).
* Long-term treatment with bisphosphonates, corticosteroids, anti-inflammatory, anticonvulsant, antiepileptics, fibrates.
* Known hypersensitivity to vitamin D
* Prior supplementation (in the last year) or supplementation of vitamin D during
* Participation at the time of inclusion in the trial, or planned participation during the same period that this trial, another trial on a vaccine, drug, medical device.
* Vaccination during the 4 weeks prior to vaccination or immunization of the test set out in the three weeks after vaccination test.
* Transfusion of immunoglobulins, blood or blood products during the last 3 months
* Congenital or acquired, known or suspected immunodeficiency, immunosuppressive therapy in the last 6 months, such as cancer chemotherapy or radiotherapy; steroids long-term systemic (prednisone or equivalent for more than two consecutive weeks in the Previous 3 months).
* Systemic Hypersensitivity to any component of the vaccine (ovalbumin, chicken protein, neomycin, formaldehyde, octoxinol 9), or a history of reaction to influenza vaccine or a vaccine containing one of the substances in the vaccine trial, which involved life-threatening.
* Deprivation of liberty or by administrative order issued by a court, subject to emergency medical or involuntary hospitalization.
* Topic enjoying a measure of legal protection (guardianship, guardianship ...).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
levels of cathelicidin | at Month 3

SECONDARY OUTCOMES:
Levels of plasma 25(OH) D | Day 0, week 7 and Month 3.
Levels of pro-inflammatory cytokines and anti-inflammatory (IL-4, IL-5, IL-10, IL-13, IL-17, IL-23, TFN, IFN and TGF) | Day 0, week 7 and Month 3.
Rate of seroconversion, seroprotection, the MGT antibodies | Day 0, week 7 and Month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Henri LAURICHESSE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Goncalves-Mendes N, Talvas J, Duale C, Guttmann A, Corbin V, Marceau G, Sapin V, Brachet P, Evrard B, Laurichesse H, Vasson MP. Impact of Vitamin D Supplementation on Influenza Vaccine Response and Immune Functions in Deficient Elderly Persons: A Randomized Placebo-Controlled Trial. Front Immunol. 2019 Feb 8;10:65. doi: 10.3389/fimmu.2019.00065. eCollection 2019. PMID 30800121